CLINICAL TRIAL: NCT01650662
Title: CYCLosporinE A in Reperfused Acute Myocardial Infarction Prospective, Controlled, Randomized, Multicentre Trial to Examine Whether a Single i.v. Bolus of Cyclosporine A Before PCI Can Reduce Myocardial Reperfusion Injury in Patients With STEMI.
Brief Title: CYCLosporinE A in Reperfused Acute Myocardial Infarction
Acronym: CYCLE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: Heart Care Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CYCLE (IRFMN_5635); 2011-002876-18 (EudraCT Number)
Record Dates: First submitted 2012-07-24; First posted 2012-07-26 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2013-10

CONDITIONS: Acute Myocardial Infarction
Keywords: Acute Myocardial Infarction; Cyclosporine A; Reperfusion; Clinical Trial
MeSH Terms: interventions — Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cyclosporine A (Experimental): The investigational active treatment is CsA, an immunosuppressant indicated for the prevention of acute rejection after organ transplant, including cardiac transplantation.
  The preparation used in the trial will be Sandimmun IV, containing CsA 50 mg/ml, Cremophor® EL and 94% ethyl alcohol in a 5 ml vial.
  Patients will received Cyclosporine A on the top of recommended standard care for acute myocardial infarction.
  Interventions: Drug: Cyclosporine A
- Control group (Experimental): The control group received on the top of recommended standard care for acute myocardial infarction.
  Interventions: Drug: Cyclosporine A

INTERVENTIONS:
Drug: Cyclosporine A — In the CsA group, at least 5 min before balloon inflation and stenting, patients will receive an intravenous bolus injection of 2.5 mg/kg of CsA. In the control group, patients will receive only recommended treatments. CsA will be dissolved in normal NaCl 0.9% solution (final concentration 25 mg/ml) and injected slowly (over 20-30 seconds) via a catheter positioned in an antecubital vein at least 5 min before PCI, to allow for distribution of the drug.

SUMMARY:
Infarct size is a major determinant of prognosis after myocardial infarction (MI). It has been reported that Cyclosporine A (CsA) administered immediately prior to percutaneous coronary intervention (PCI) significantly could reduce reperfusion injury and consequently infarct size in ST elevation MI (STEMI) patients.

CYCLE trial is a multicenter, controlled, randomized open label study, with blind assessment of endpoint measures. The objective is to determine whether a single i.v. dose of CsA within 6 hour onset of symptoms of STEMI in 444 patients, improves outcomes after successful primary PCI, by reducing myocardial injury associated to reperfusion.

DETAILED DESCRIPTION:
The possibility of optimizing the results of an early and effective reopening of the occluded artery by reducing/avoiding the impact of the so-called reperfusion injury has been for many years one of the most elusive objectives of pharmacological research, with evolving hypothesis and targets.

A recently published trial has provided support to a line of investigation focused on the role of mitochondrial dysfunction, the so-called permeability transition, as cause of irreversible myocardial injury associated to reperfusion. In fact, a single dose of the widely used immunosuppressant agent, CsA, a potent inhibitor of mitochondrial permeability transition pore opening, was reported to limit ischemia-reperfusion injury in 50 patients with anterior MI who underwent primary PCI.

Since infarct size and left ventricular function are the main determinants of long-term morbidity and mortality, a single measure to limit infarct size is of potential clinical benefit. Therefore the results of the previously mentioned trial should be replicated in a larger sample size, before going on to a trial with clinical endpoints.

- Sample size

Assuming an incidence of the primary endpoint of 55% in the control group, we calculated that 444 patients (222 patients per group) will be required for the study to have 80% power to detect a 25% relative improvement (resulting in an endpoint frequency of 68.7% in the CsA group) with a 5% drop-out rate and a two-sided alpha level of 5%. The size of the trial will allow to investigate treatment benefit for the secondary endpoint hsTnT: assuming a concentration of 2.7 ng/mL on day 4 (common SD=2.1) in the control group, the study will have a 90% power to show a 25% reduction with CsA at a two-sided alpha level of 5%.

- Safety

Adverse events with intravenous CsA (i.e. anaphylactoid reactions/anaphylactic shock, acute renal failure, or hypertensive crisis) are reported to be very rare. In this trial, patients will receive only one iv dose of CsA, therefore we expect a low probability of adverse effects related to repeated administrations, i.e. acute renal failure or hypertensive crisis. Nonetheless a close monitoring of the safety of the single dose of CsA is foreseen with monthly examination of data of safety by the Steering Committee.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with large STEMI not older than 6 hours, defined as
* angina pectoris or equivalent symptoms of more than 20 minutes duration within last 6 hours, and
* ST elevation in at least 3 leads in anterior MI and/or a deviation in at least 4 leads in inferior MI,
* TIMI flow 0 or 1 in identified culprit artery
* Intended acute primary PCI
* Age ≥ 18 years
* Ability to understand the nature, scope, and possible consequences of the study participation/legal capacity
* Written informed consent

Exclusion Criteria:

* Left bundle branch block
* TIMI flow > 1 in the identified culprit artery
* Treatment with CsA within last 10 days
* Contraindication to CsA or history of allergic reaction to CsA
* Coronary anatomy not suitable for PCI
* Thrombolytic therapy within 24 h. before randomization
* Previous MI
* Previous CABG
* Severe renal or hepatic insufficiency
* Malignant tumor, not curatively treated
* Women with childbearing potential, esp. pregnant or nursing women
* Participation in another clinical or device trial within the previous 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2012-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Improvement of myocardial reperfusion, measured with ST-segment resolution >=70% | 1 hour after percutaneous coronary intervention (PCI)
  Improvement of myocardial reperfusion, measured with ST-segment resolution >=70% 1 hour after PCI

SECONDARY OUTCOMES:
High sensitive cardiac troponin T (hs-cTnt). | at day 4 after percutaneous coronary intervention (PCI)
  High sensitive cardiac troponin T (hs-cTnt) at day 4 after PCI; ; this will be the most relevant among secondary endpoints given its value as readout of cardiac protection.
Clinical events: all-cause mortality, HF or shock; rehospitalization for CV reasons | within 6 months of randomization
  Clinical events within 6 months of randomization: all-cause mortality, HF or shock; rehospitalization for CV reasons.
Infarct size: Troponin curve (T or I, assayed locally) | Time course of troponin release during the first 72 hours after the visualization of the antegrade flow.
  Infarct size: Troponin curve (T or I, assayed locally); The time course of troponin release during the first 72 hours after the visualization of the antegrade flow, will be studied.
LV remodeling and function as assessed by echocardiography; | at 6 months after randomization
  LV remodeling and function at 6 months, as assessed by echocardiography;
No reflow, as assessed by myocardial blush | 1 day (after the visualization of the antegrade flow)
  No reflow, as assessed by myocardial blush after the visualization of the antegrade flow

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Latini, MD, Study Chair — Mario Negri Institute, Milan, Italy; Filippo Ottani, MD, Study Chair — Ospedale G.B. Morgagni, Pierantoni, Forlì, Italy
Locations (31):
- Italy (31):
  - Ospedale Regionale Umberto Parini, Aosta, AO
  - Ospedale S. Donato, Arezzo, AR
  - Ospedale San Paolo, Bari, BA
  - Azienda Ospedaliera di Seriate, Seriate, BG
  - Azienda Ospedaliera di Treviglio, Treviglio, BG
  - Policlinico S.Marco, Zingonia - Osio Sotto, BG
  - Ospedale Maggiore, Bologna, BO
  - Istituto Fondazione Poliambulanza, Brescia, BS
  - Azienda Ospedaliera G.Brotzu, Cagliari, CA
  - Azienda Ospedaliera Santa Croce e Carle, Cuneo, CN
  - Ospedale G.B. Morgani - L. Pierantoni, Forlì, Forli
  - Ospedale delle Misericordie, Grosseto, GR
  - Ospedale Campo di Marte, Lucca, LU
  - Ospedale di Desio, Desio, MB
  - Policlinico Monza, Monza, MB
  - AOR Villa Sofia - Cervello P.O., Palermo, PA
  - AOR Villa Sofia - Cervello PO Villa Sofia, Palermo, PA
  - Ospedale Civile dello Spirito Santo, Pescara, PE
  - Ospedale Santa Maria delle Croci, Ravenna, RA
  - Ospedale San Camillo, Roma, RM
  - Ospedale Infermi, Rimini, RN
  - Ospedale Santa Corona, Pietra Ligure, SV
  - Ospedale Santa Chiara, Trento, TN
  - Ospedale degli Infermi, Rivoli, TO
  - Ospedale Maria Vittoria, Torino, TO
  - Azienda Ospedaliera Universitaria - Ospedale Riuniti, Trieste, TS
  - Ospedale S. Giacomo, Castelfranco Veneto, TV
  - Ospedale Ca' Foncello, Treviso, TV
  - Azienda Ospedaliera -Univ. S. Maria delle Misericordie, Udine, UD
  - Ospedale dell'Angelo, Mestre, VE
  - Ospedale Civile San Bortolo, Vicenza, VI

REFERENCES:
- [Derived] Ottani F, Latini R, Staszewsky L, La Vecchia L, Locuratolo N, Sicuro M, Masson S, Barlera S, Milani V, Lombardi M, Costalunga A, Mollichelli N, Santarelli A, De Cesare N, Sganzerla P, Boi A, Maggioni AP, Limbruno U; CYCLE Investigators. Cyclosporine A in Reperfused Myocardial Infarction: The Multicenter, Controlled, Open-Label CYCLE Trial. J Am Coll Cardiol. 2016 Feb 2;67(4):365-374. doi: 10.1016/j.jacc.2015.10.081. PMID 26821623
- See also: The protocol presentation, can be found in the window of CYCLE Study. — http://www.anmco.it